CLINICAL TRIAL: NCT00001569
Title: Phase I Trial of Continuous Hyperthermic Peritoneal Perfusion (CHPP) With Cisplatin Plus Early Postoperative Intraperitoneal Paclitaxel and 5-FU for Peritoneal Carcinomatosis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 970072; 97-C-0072
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2002-12

CONDITIONS: Carcinoma; Peritoneal Neoplasm
Keywords: Gastrointestinal; Adenocarcinoma; Taxol
MeSH Terms: conditions — Carcinoma; Peritoneal Neoplasms; Adenocarcinoma | interventions — Cisplatin; Paclitaxel; Fluorouracil

INTERVENTIONS:
Drug: Cisplatin
Drug: Paclitaxel
Drug: 5-FU

SUMMARY:
Two days prior to planned surgery, paclitaxel is infused IV over 24 hours.

Patients will undergo cytoreductive surgery, to debulk tumor. Scope of procedure will vary with each patient, including a spectrum of possible procedures, such as splenectomy, liver resection, pancreatic resection or bowel resection.

After cytoreductive surgery, continuous hyperthermic peritoneal perfusion (CHPP) surgery with cisplatin will begin by placing an influx and efflux catheters via abdominal wall. Perfusion rate of cisplatin is 1.5 L/min and the duration is 90 min.

Postoperative intraperitoneal chemotherapy will begin 24 hours after CHPP surgery.

Dose escalation will proceed after patients at a given dose level receive 3 courses. In order to properly evaluate hematoxicity, a minimum of 3 weeks will be required before dose escalation. MTD is either the dose level immediately below the level at which 2 of 6 patients in a cohort experience nonhematologic dose limiting toxicity (DLT) or when 4 of 6 patients experience hematologic DLT.

Two to 4 months after surgery, laparotomy will be conducted to determine response to treatment. If tumor size is decreased, patients will undergo a second treatment course identical to the same techniques and chemotherapy agents.

DETAILED DESCRIPTION:
Peritoneal carcinomatosis is considered a terminal stage of tumor progression. Cytoreductive surgery plus aggressive combination intraperitoneal chemotherapy may significantly alter the natural history of this disease. This study will define the maximum tolerated dose of paclitaxel and 5-fluorouracil (5-FU) given as an early post-operative intraperitoneal (IP) dwell therapy after cytoreductive surgery and continuous hyperthermic peritoneal perfusion with cisplatin (CHPP).

ELIGIBILITY:
The patients must have an ECOG performance status of 0 or 1 and have no concomitant medical problems that would place them at increased risk for a major surgical procedure (EG, cardiac or pulmonary disabilities).

Patients at increased risk for coronary artery disease or cardiac dysfunction (e.g., age greater than 65, history of hypertension, first degree relative with atherosclerotic coronary artery disease) will undergo cardiac evaluation and performed which will include an attempt to remove all disease greater than 0.5 cm in diameter.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 74
Dates: Start 1997-01; Study Completion 2002-12

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Institute (NCI), Bethesda, Maryland, United States

REFERENCES:
- [Background] Fujimoto S, Shrestha RD, Kokubun M, Ohta M, Takahashi M, Kobayashi K, Kiuchi S, Okui K, Miyoshi T, Arimizu N, et al. Intraperitoneal hyperthermic perfusion combined with surgery effective for gastric cancer patients with peritoneal seeding. Ann Surg. 1988 Jul;208(1):36-41. doi: 10.1097/00000658-198807000-00005. PMID 3133994
- [Background] Sugarbaker PH, Gianola FJ, Speyer JC, Wesley R, Barofsky I, Meyers CE. Prospective, randomized trial of intravenous versus intraperitoneal 5-fluorouracil in patients with advanced primary colon or rectal cancer. Surgery. 1985 Sep;98(3):414-22. PMID 3898450
- [Background] Dedrick RL, Myers CE, Bungay PM, DeVita VT Jr. Pharmacokinetic rationale for peritoneal drug administration in the treatment of ovarian cancer. Cancer Treat Rep. 1978 Jan;62(1):1-11. PMID 626987